CLINICAL TRIAL: NCT06036758
Title: VIDAS® NEPHROCLEAR CCL14 Diagnostic Accuracy Study
Brief Title: VIDAS® NEPHROCLEAR Diagnostic Accuracy Study
Status: Completed | Type: Observational
Sponsor: BioMérieux (Industry)
Responsible Party: Sponsor
Other Study IDs: B3166-CTPR02
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-09

CONDITIONS: Acute Kidney Injury; Stage 2 Acute Kidney Injury; Stage 3 Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Persons with Stage 2 to Stage 3 AKI: Persons with Stage 2 to Stage 3 AKI who are in the ICU.
  Interventions: Diagnostic Test: VIDAS® NEPHROCLEAR™ CCL14 Test

INTERVENTIONS:
Diagnostic Test: VIDAS® NEPHROCLEAR™ CCL14 Test — Urine samples previously collected from persons with stage 2/stage 3 AKI will be tested using the VIDAS® NEPHROCLEAR™ CCL14 Test

SUMMARY:
This is a multi-center sample analysis study in which urine samples previously collected from persons with Stage 2 or Stage 3 Acute Kidney Injury (AKI), will be tested in order to validate the VIDAS® NEPHROCLEAR™ CCL14 Test

DETAILED DESCRIPTION:
The VIDAS® NEPHROCLEAR™ CCL14 Test is intended to be used in conjunction with clinical evaluation, in ICU patients with moderate to severe (stage 2 or 3) acute kidney injury (AKI), as an aid in the risk assessment for developing persistent severe AKI (stage 3 AKI lasting ≥ 72 hours) within 48 hours of patient assessment.

The VIDAS® NEPHROCLEAR™ CCL14 Test is intended to be used in patients 21 years of age or older.

The objective of this study is to evaluate the diagnostic accuracy of the VIDAS® NEPHROCLEAR™ CCL14 test when used on the VIDAS® 3 instrument. Sensitivity, specificity, negative predictive value (NPV), positive predictive value (PPV), likelihood ratios (LR), and relative risk (RR), will be evaluated at the pre-determined cut-off values.

Previously collected urine samples from persons with Stage 2 to Stage 3 AKI will be tested in this study. The VIDAS® test results will be compared to the clinical AKI status established by independent adjudication by medical professionals, that are blinded to the VIDAS® test results.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 21 years of age or older;
* Receiving care in an intensive care unit;
* Expected to remain in the ICU for at least 48 hours after enrollment;
* Use of indwelling urinary catheter as standard care at the time of enrollment;
* Subject must have acute kidney injury (KDIGO Stage 2 or Stage 3) at the time of sample collection;
* Urine sample must be collected within 36 hours of meeting KDIGO Stage 2 criteria;
* Documented informed consent provided by patient or legally authorized representative (LAR).

Exclusion Criteria:

* Prior kidney transplantation;
* Comfort-measures-only status;
* Already receiving dialysis (either acute or chronic) or in imminent need of dialysis at the time of enrollment;
* Known infection with human immunodeficiency virus (HIV) or active hepatitis (acute or chronic); (NOTE: HIV or hepatitis testing need not be performed for enrollment in this study.)
* Special populations, pregnant women, prisoners or institutionalized individuals;

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with Stage 2 to Stage 3 AKI
Sampling Method: Non-Probability Sample
Enrollment: 477 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Risk of developing persistent severe AKI | Within 48 hours of ICU admittance
  The urine sample collected from ICU patients will be tested using the VIDAS® NEPHROCLEAR™ CCL14 Test, which is intended to be used in conjunction with clinical evaluation, in ICU patients with moderate to severe (stage 2 or 3) acute kidney injury (AKI), as an aid in the risk assessment for developing persistent severe AKI (stage 3 AKI lasting ≥ 72 hours) within 48 hours of patient assessment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - George Washington University, Washington D.C., District of Columbia
  - University of Illinois, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No